CLINICAL TRIAL: NCT03938506
Title: The Assessment of the Pilot Balloon Palpation Method in Different-sized Endotracheal Tubes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2019-0104
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Intubation, Intratracheal
Keywords: Adult male patients who require endotracheal intubation using the endotracheal tube size of 6.0 or 8.0; endotracheal tube cuff

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intubation using the endotracheal tube size of 6.0 or 8.0: Adult male patients who require endotracheal intubation using the endotracheal tube size of 6.0 or 8.0
  Interventions: Other: cuff pressure of the endotracheal tube

INTERVENTIONS:
Other: cuff pressure of the endotracheal tube — The endotracheal intubation will be performed after the anesthetic induction. The cuff will be inflated using the air by the palpation method. The cuff pressure of the endotracheal tube will be measured using the manometer.

SUMMARY:
Endotracheal tube is a commonly used for general anesthesia in head and neck surgery. It is necessary to place the endotracheal tube in the trachea of the patient and then inflate the cuff with air. This is because the air-inflated cuff contacts the inner wall of the patient's trachea to deliver oxygen through the tube. If the cuff does not inflate, oxygen will leak through the space between the cuff and the patient's trachea. In addition, the risk of pneumonia increases. Therefore, after placing the endotracheal tube in the patient's trachea, the cuff is immediately inflated with air. However, when the cuff is inflated using an excess of air, the cuff may pressurize the mucous membrane of the tracheal wall and cause ischemia. Pressure in the over-inflated cuff was also found to be associated with post-operative sore throat, vocal cord paralysis, and nerve damage. Therefore, appropriate amount of air should be used to inflate the cuff into the air and adjust the pressure within the cuff to be within the range of 20-30 cmH2O. The common method to inflate the endotracheal tube cuff is palpation method. However, the palpation of the cuff is not accurate because of the different size between the pilot balloon and the cuff. Thus, the investigators hypothesized that the different size of the tube will affect the accuracy of the palpation method.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult male patients who require endotracheal intubation using the endotracheal tube size of 6.0 or 8.0

Exclusion Criteria:

* 1. Patients under 20 years old
* 2. Patients receiving emergency surgery
* 3. Patients with tracheostomy tubes
* 4. Pregnant women
* 5. Patients who can not read the consent form or are not fluent in Korean
* 6. Patients who refused the clinical trial
* 7. Patient with endotracheal mass in the trachea where the cuff is located
* 8. Tracheal deviation is observed in the neck due to tumor in the neck

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male patients who require endotracheal intubation using the endotracheal tube size of 6.0 or 8.0
Sampling Method: Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
The incidence rate when the pressure in the cuff of the endotracheal tube is not within the proper range. | participants will followed until the completion of the anesthetic induction (less than 15 minutes).
  the investigator will monitor the pressure of the endotracheal tube cuff after anesthetic induction.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Ban MG, Kim SY, Kim MS, Park WK, Kwon YI, Kim HJ. Accuracy of pilot balloon palpation for cuff pressure assessment in small versus large sized tubes: a prospective non-randomized observational study. Sci Rep. 2023 Apr 5;13(1):5580. doi: 10.1038/s41598-023-32704-3. PMID 37020098